CLINICAL TRIAL: NCT01498523
Title: An Explorative Study to Characterize the Glycaemic and Insulinaemic Responses of Regular Camel Milk and Camel Milk Powder
Brief Title: The Glycaemic and Insulinaemic Responses of Camel Milk
Acronym: GLUCAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 38520
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Camel milk; Postprandial glycaemic response; postprandial insulinaemic response; Glycaemic index

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- raw camel milk (Experimental)
  Interventions: Other: Camel milk
- camel milk powder solution (Experimental)
  Interventions: Other: camel milk powder solution
- raw cow milk (Active Comparator)
  Interventions: Other: raw cow milk
- Glucose solution (Active Comparator)
  Interventions: Other: Glucose solution

INTERVENTIONS:
Other: Camel milk — 600ml of raw camel milk will be consumed in 10 minutes. the blood glucose concentrations will be measured at 0, 15, 30, 45, 60 ,90 and 120 minutes by finger-prick blood samples. Also, blood insulin and amino acids concentration will be measured at 0, 30 and 75 minutes.
  Other Names: Dromedary milk
  Arms: raw camel milk
Other: camel milk powder solution — 72g camel milk powder will be dissolved in 540ml water to make 600ml camel milk powder solution. This will be consumed in 10 minutes. the blood glucose concentrations will be measured at 0, 15, 30, 45, 60 ,90 and 120 minutes by finger-prick blood samples. Also, blood insulin and amino acids concentration will be measured at 0, 30 and 75 minutes.
  Other Names: Dromedary milk powder
  Arms: camel milk powder solution
Other: raw cow milk — 50ml water will be added to 550ml raw cow milk to make 600ml cow milk. This will be consumed in 10 minutes. the blood glucose concentrations will be measured at 0, 15, 30, 45, 60 ,90 and 120 minutes by finger-prick blood samples. Also, blood insulin and amino acids concentration will be measured at 0, 30 and 75 minutes.
  Other Names: Bovine milk
  Arms: raw cow milk
Other: Glucose solution — 25g glucose will be dissolved in 600ml water, and this will be consumed in 10 minutes. the blood glucose concentrations will be measured at 0, 15, 30, 45, 60 ,90 and 120 minutes by finger-prick blood samples. Also, blood insulin and amino acids concentration will be measured at 0, 30 and 75 minutes.
  Other Names: Sugar solution
  Arms: Glucose solution

SUMMARY:
Rationale: Recently, human, animal and epidemiological studies suggested that camel milk has a hypoglycaemic activity. However, a mechanism and reasons for this activity have not been sufficiently studied. Therefore, a study on a glycaemic and insulinaemic responses of regular camel milk and camel milk powder is needed.

Objective: To explore the glycaemic and insulinaemic responses of regular camel milk and camel milk powder in healthy adults.

Study design: In a randomised, single-blind and cross over design, two hour post prandial glucose and insulin responses of 4 treatments (regular camel milk, camel milk powder, regular cow milk and glucose) will be measured . Those treatments will be consumed in a portion that contained 25g available carbohydrate. Finger-prick capillary blood samples will be taken at fasting, and 15, 30, 45, 60, 90, 120 minutes after ingestion of the test product. Venepunctures will be taken at fasting, 30 and 75 minutes after ingestion of the test product. The measurements will be conducted on 4 separate days with at least 2 days wash out.

Study population: 20 healthy volunteers aged 18 to 35 years, with BMI between 18.5 to 25 kg/m2.

Intervention: The treatments are regular camel milk, camel milk powder, regular cow milk and glucose. These are standardized to 600ml containing 25g available carbohydrate.

Main study parameters/endpoints: Main parameters are postprandial blood glucose and insulin responses. Secondary parameters: amino acid composition and glycemic index.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This intervention is non-therapeutic to the subjects. The risk associated with participation is negligible and the burden can be considered low. Before subjects are able to participate in this study they will have to fill out a brief questionnaire, and have their fasting blood glucose measured, in order to ensure they fit the inclusion criteria of the study. Once entering the study, each subject will have to visit the research centre 4 times for the postprandial tests. On each measurement day, each subject will be required to have fasted for at least ten hours before (an overnight fast). Each subject will have 7 finger-prick blood samples and 3 venapunctures taken during each visit. A maximum amount of 50 ml blood is drawn per day.

DETAILED DESCRIPTION:
There is no detailed description

ELIGIBILITY:
Inclusion Criteria:

* Healthy: as judged by the subjects;
* Age: 18 to 35.

Exclusion Criteria:

* Pregnant or lactating females;
* Presence of a chronic disease such as diabetes, illness, dysmetabolic syndrome;
* 18.5 > BMI > 25 kg/m2;
* Lactose intolerance or experiencing discomfort after milk consumption;
* Weight loss or gain of more than 5 kg in the last two months;
* Using an energy restricted diet during the last 2 months;
* Fasting blood glucose levels >100 mg/dl or 5.6 mmol/l (18);
* Smokers;
* Use of medications other than birth control, paracetamol, aspirin, asthma or hay fever;
* Previous problems with blood sampling.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
blood glucose and insuline concentrations | 2 months
  During the test session, subjects will drink raw camel milk, camel milk powder solution, raw cow milk and glucose solution. At time points 0, 15, 30, 45, 60, 90 and 120 minutes blood glucose level will be measured by finger-prick blood samples. Also, at time points 0, 30, 75 minutes insulin level will be measured by venepuncture blood samples.

SECONDARY OUTCOMES:
Blood amino acids concentration | 2 months
  During the test session, subjects will drink raw camel milk, camel milk powder solution, raw cow milk and glucose solution. At time points 0, 30, 75 minutes blood amino acids level will be measured by venepuncture blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Feskens, Prof.Dr.Ir., Study Director — Wageningen University; Anne Wanders, MSc, Principal Investigator — Wageningen University; Monique van Nielen, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands